CLINICAL TRIAL: NCT06324721
Title: The Enigma of Subjective Lymphedema: Who and Why do Patients Report Lymphedema After Breast Cancer Treatment Without an Objective Measurable Swelling? The Role of Lymphatic and Sensory Processing Problems
Brief Title: Who and Why do Patients Report Lymphedema After Breast Cancer Treatment Without an Objective Measurable Swelling
Acronym: LymphSens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Nele Devoogdt, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: S68133
Record Dates: First submitted 2024-03-12; First posted 2024-03-22 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Lymphedema; Sensory Processing Disorder
Keywords: lymphedema; subclinical edema; nociceptive problems; neuropathic problems; central sensory problems
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Weights and Measures; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients (Experimental): Women and men who are being diagnosed with primary unilateral non-metastatic or oligometastatic breast cancer and scheduled for breast surgery in combination with axillary lymph node dissection or sentinel node biopsy
  Interventions: Other: Measurements for breast cancer related lymphedema (volumetric measurements, bioimpedance spectroscopy, bioimpedance analysis, tissue dielectric constant measurements, ultrasonography); Other: Measurements for lymphatic problems (volumetric measurements, tissue dielectric measurement, lymphofluoroscopy); Other: Measurements for sensory processing problems by monofilaments, algometer, goniometer, and neurosensory analyzer

INTERVENTIONS:
Other: Measurements for breast cancer related lymphedema (volumetric measurements, bioimpedance spectroscopy, bioimpedance analysis, tissue dielectric constant measurements, ultrasonography) — Assessments related to different types of breast cancer related lymphedema at arm (1. self-reported swelling at arm, 2. subjective arm lymphedema, 3. objective arm lymphedema) using the Norman questionnaire, volume measurements (volumetry and perimetry), bioimpedance spectroscopy, and bioimpedance analysis
  Assessments related to different types of breast cancer related lymphedema at trunk/ breast (1. self-reported swelling at trunk/ breast, 2. subjective trunk/ breast lymphedema, 3. objective trunk/ breast lymphedema) using the Norman questionnaire, tissue dielectric measurements, and ultrasonography
Other: Measurements for lymphatic problems (volumetric measurements, tissue dielectric measurement, lymphofluoroscopy) — Clinical assessments related to lymphatic problems (1. amount of swelling at arm by relative arm volume difference, 2. amount of swelling at trunk by percentage water ratio, 3. severity of dermal rerouting at upper limb and trunk by lymphofluoroscopy (i.e., near-infrared fluorescence imaging device)
Other: Measurements for sensory processing problems by monofilaments, algometer, goniometer, and neurosensory analyzer — Clinical measurements related to nociceptive, neuropathic and central sensory problems based on the Quantitative Sensory Testing principles using different devices algometer, goniometer, standardized set of monofilaments, and neurosensory analyzer

SUMMARY:
Breast cancer related lymphedema (BCRL) at the arm and/or trunk is an extremely dreaded complication after breast cancer treatment due to its chronicity and impact.

The incidence of objective arm and trunk/ breast BCRL is declining due to the major shift into the treatment approach of breast cancer. However, many patients report a sensation of swelling without the presence of objective BCRL, referred to as subjective BCRL. Therefore, subjective BCRL is defined as the diagnosis of BCRL based on the patient's sensation of a difference in size at the arm and/or trunk without the presence of objective BCRL.

At this moment, there is no clear information on the prevalence and the transitions between different BCRL states (no-subjective-objective) over time, as well as about the underlying mechanisms and contributing factors of subjective BCRL. Therefore, the investigators hypothesize that four mechanisms might be associated with the presence and severity of subjective arm or trunk/breast BCRL, including the presence and/ or severity of lymphatic (1) and sensory processing problems (nociceptive (2), neuropathic (3), and/or central sensory processing problems (4)).

The investigators will set up a prospective longitudinal study with breast cancer patients to determine the prevalence of subjective and objective arm or trunk/ breast BCRL at 1, 6, and 12 month(s) post-surgery and the transitions between different BCRL states (no-subjective-objective BCRL) (AIM 1). In addition, factors related to four potential underlying mechanisms (lymphatic, nociceptive, neuropathic, and central sensory processing problems) that contribute to the occurrence of subjective BCRL in comparison to no self-reported swelling and objective BCRL will be determined (AIM 2). Furthermore, the present study will be undertaken to determine factors related to these four underlying mechanisms that contribute to the severity of subjective BCRL at arm or trunk/ breast BCRL within the group of patients with subjective BCRL at different time-points after surgery (at 1, 6, and 12 month(s) post-surgery) (AIM 3).

ELIGIBILITY:
Inclusion criteria:

1. adults (men and women) who are ≥ 18 years of age
2. diagnosed with primary unilateral non-metastatic or oligometastatic breast cancer
3. scheduled for surgery (mastectomy or breast conserving surgery; in combination with axillary lymph node dissection or sentinel node biopsy)
4. able to read, understand, and speak Dutch
5. have voluntary written informed consent of the patient

Exclusion Criteria:

1. distant metastases
2. planned bilateral lymph node surgery
3. oedema of the arm from another cause
4. an allergy to iodine or Indocyanine Green (ICG), or
5. physically or mentally unable to participate throughout the entire duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Presence of subjective arm lymphedema | Time frame up to 12 months post-surgery
  The presence of subjective arm lymphedema will be determined by the combination of two items.
  If self-reported swelling at arm is "yes" and objective arm BCRL is "no", then the presence of subjective arm BCRL will be defined as yes.
  To determine the presence of self-reported swelling at arm, we will use the Norman Questionnaire. If the patient responds ''yes'' to the item self-reported difference in the sizes of at least one of 3 sites (hand, lower arm, and upper arm), the presence of 'self-reported swelling at arm' is recorded as ''yes''.
  To determine the presence of objective lymphedema at arm, please see outcome 3.
  Unit of the outcome measure is yes/no.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Presence of subjective trunk/ breast lymphedema | Time frame up to 12 months post-surgery
  The presence of subjective trunk/ breast lymphedema will be determined by the combination of two items.
  If self-reported swelling at trunk/ breast is "yes" and objective trunk/ breast BCRL is "no", then the presence of subjective trunk/ breast BCRL will be defined as yes.
  To determine the presence of self-reported swelling at trunk/ breast, we will use the Norman Questionnaire. If the response is ''yes'' to the item self-reported difference in the sizes of at least one of these 2 sites (trunk or breast region), the presence of ''self-reported swelling in the trunk/breast'' is recorded as ''yes.''
  Unit of the outcome measure is yes/no.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Presence of objective arm lymphedema | Time frame up to 12 months post-surgery
  4 methods are used to determine the presence of objective arm lymphedema: a) relative hand volume difference, b) relative arm volume difference, c) bioimpedance analysis, and d) bioimpedance spectroscopy at arm region
  If at least one of four cut-off values is present, the presence of objective arm lymphedema will be considered as yes:
  1. an increase of relative hand volume difference between the affected and non-affected hands of ≥5% compared to the baseline difference OR
  2. an increase of relative arm volume difference between the affected and non-affected arms of ≥5% compared to the baseline difference OR
  3. Extra-cellular water ratio by Bioimpedance Analysis at affected arm of >0.3850 OR
  4. Extracellular water ratio by Bioimpedance Spectroscopy, >6.5 change in the L-Dex score from the baseline score
  Unit of the outcome measure is yes/no.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Presence of objective trunk/ breast lymphedema | Time frame up to 12 months post-surgery
  2 methods are used to determine the presence of objective trunk/breast lymphedema: a) tissue dielectric measurement, b) skin thickness measurement at trunk/breast region
  If one of four criteria is present, the presence of objective trunk/ breast lymphedema will be considered as yes:
  1. percentage of water content ratio at the trunk ≥ 1.32 OR
  2. percentage of water content ratio at the trunk ≥ 1.40 OR
  3. > 2 standard deviations (SD) from the average skin thickness in at least one reference point on the trunk compared to the reference value at pre-surgery OR
  4. > 2 SD from the average skin thickness in at least one reference point one quadrant of the affected breast compared to the reference value at pre-surgery
  Unit of the outcome measure is yes/no.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery

SECONDARY OUTCOMES:
Amount of swelling at upper limb and trunk/breast | Time frame up to 12 months post-surgery
  See outcomes 3 and 4 Presence of objective arm and trunk/ breast BCRL Total upper limb (hand + arm) volume is calculated by taking the sum of the hand volume and relative arm volume. Then, the difference between both upper limb is calculated. Relative upper limb volume difference is used for analysis.
  Average percentage water (PWC) value of reference points is calculated. PWC ratio=PWC affected side at post-surgery/PWC reference value at baseline is used for analysis.
  Assessment at pre-surgery, 1 month, 6 months, and 12 months post-surgery
Severity of dermal rerouting at upper limb and trunk/breast | Time frame up to 12 months post-surgery
  Lymphofluoroscopy will be used. Indocyanine green (ICG)/ aqua is injected in the patient's hand; linear (normal) and dermal rerouting patterns are visualized after 90 minutes of the injection. The body is divided into 14 areas (11 areas at upper limb and 3 areas at trunk/breast). Each area is scored between 0 and 3: 0 (normal pattern), 1 (splash pattern), 2 (stardust pattern), and 3 (diffuse pattern).
  Total dermal rerouting score for arm is between 0 and 33. Total dermal rerouting score for trunk/ breast is between 0 and 9.
  Assessment at 1 month, 6 months, and 12 months post-surgery
Severity of myofascial adhesions at the level of the scars | Time frame up to 12 months post-surgery
  The evaluation tool for Myofascial Adhesions in Patients after Breast Cancer (MAP-BC evaluation tool): assessed at 2 locations (i.e., axillary scar and breast or mastectomy scar). Each location is palpated for adhesions at 3 levels (i.e., skin, superficial, and deep) on a 4-points scale (0- no restriction, 1-limited restriction, 2-early and hard restriction, and 3-very stiff and tissue gliding is not possible). The total score of the MAP-BC is calculated by taking the sum of each item and is used for the analysis
  Total score ranges between 0 - 18.
  Assessment at 1 month, 6 months, and 12 months post-surgery
Severity of local muscle stiffness | Time frame up to 12 months post-surgery
  Myofascial tissue stiffness will be evaluated at the affected and non-affected sides of the pectoralis major, infraspinatus, and teres major muscles.
  Average muscle stiffness score of 3 muscles at affected and non-affected side is calculated.
  Then, the local muscle stiffness ratio is calculated: Average muscle stiffness at the affected side in N/m/Average muscle stiffness at the non-affected side and this ratio is used for the analysis.
  Unit of the outcome measure is Newton/ meter.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of local muscle tenderness | Time frame up to 12 months post-surgery
  Pressure pain thresholds will be evaluated using digital algometer on affected and non-affected sides of pectoralis major, infraspinatus, and teres major muscles. Increasing pressure (1kg/sec) is applied perpendicularly to the skin. Patient is asked to say 'stop' when the sensation of pressure first changes to unpleasant feeling. 2 measurements are taken at each reference point.
  Average pressure pain thresholds of 2 measurements at affected and non-affected side is calculated. The local muscle tenderness ratio is calculated: Average pressure pain thresholds at the affected side/ average pressure pain thresholds at the non-affected side and this ratio is used for the analysis.
  Unit of the outcome measure is kilogram per square centimeter (kg/cm2).
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of impaired shoulder range of motion | Time frame up to 12 months post-surgery
  Arm abduction range is evaluated by the digital goniometer. Patient is instructed to perform one shoulder abduction movement with full elbow extension and neutral wrist flexion/extension in the standing position.
  Ratio of affected shoulder abduction range of motion/non-affected shoulder abduction range of motion is calculated and used for the analysis.
  Unit of the outcome measure is degree.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Presence of neuropathic pain at upper arm and trunk | Time frame up to 12 months post-surgery
  The presence of neuropathic pain at upper arm and trunk will be evaluated by the Douleur neuropathique en 4 questions (DN4). DN4 consists of interview and examination parts. Interview part: seven items about pain descriptors. Examination part: three items about the hypoesthesia to touch and pinprick, and the presence of hyper-esthesia by the application of brushing.
  Total score ranges between 0 - 10.
  The presence of neuropathic pain is "yes" if the total score of DN4 is ≥4 .
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of sensory loss at the arm and trunk | Time frame up to 12 months post-surgery
  Mechanical detection thresholds will be determined by using standardized set of 12 nylon monofilaments at affected inner upper arm and lateral trunk. Mechanical detection threshold is defined as the lowest mechanical force identified by the patient and determined based on the principles of the Quantitative Sensory Testing. Two measurements are obtained at the affected inner upper arm and the lateral trunk. Geometric mean of the first and second detected stimulus is obtained for each location and used for the analysis.
  Average mechanical detection threshold score is between 0.25 - 512 millinewton (mN).
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of altered cold sensation sensitivity at the arm and trunk | Time frame up to 12 months post-surgery
  Cold sensation sensitivity is assessed by the Thermotest device (TSA-2 Neurosensory Analyser) at affected inner upper arm and lateral trunk. The patient pushes the button when she/he experiences a change from a thermo-neutral state to a distinct cold sensation. 3 repetitions are obtained. Average score for cold sensation sensitivity is calculated from all measurements at each assessment location.
  Unit of the outcome measure is centigrade degree.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of altered heat sensation sensitivity at the arm and trunk | Time frame up to 12 months post-surgery
  Heat sensation sensitivity is assessed by the Thermotest device (TSA-2 Neurosensory Analyser) at affected inner upper arm and lateral trunk. The patient pushes the button when she/he experiences a change from a thermo-neutral state to a distinct heat sensation. 3 repetitions are obtained. Average score for heat sensation sensitivity is calculated from all measurements at each assessment location.
  Unit of the outcome measure is centigrade degree.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of altered sensory acuity in the arm and trunk | Time frame up to 12 months post-surgery
  Sensory acuity will be evaluated using aesthesiometer at the affected inner side of upper arm and lateral side of the trunk. A stimulus is given with one or two pins on the skin of the inner side of affected upper arm and lateral side of the trunk. Patient indicates whether she/he feels one or two points. Average score of two measurements is calculated.
  Score is between 0 - 100 millimeter.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of widespread hyperalgesia | Time frame up to 12 months post-surgery
  Heat pain threshold is assessed by the Thermotest device (TSA-2 Neurosensory Analyser). Heat pain threshold is measured on the affected side at the inner upper arm and lateral trunk, and on the non-affected side at the tibialis anterior. The patient presses a button when the heat sensation is first perceived as unpleasant. 3 measurements are obtained, and the average heat pain threshold score is calculated for each assessment location. A normalized ratio is then calculated, with a higher ratio indicating decreased severity of widespread hyperalgesia.
  Normalized ratio=heat pain threshold at tibialis anterior/heat pain threshold at upper arm Normalized ratio=heat pain threshold at tibialis anterior/heat pain threshold at lateral trunk
  Unit of the outcome measure is centigrade degree.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery.
Efficacy of inhibitory pain mechanism | Time frame up to 12 months post-surgery
  A cold pressure test is performed to test the efficacy of inhibitory pain mechanism.
  The test (pressure pain threshold on the non-affected tibialis anterior muscle) and conditioning stimulus (cold stimulus on non-affected hand) is applied.
  The non-affected hand is immersed in a cold water bath of 12 centigrade degree for 60 seconds. 30 and 60 seconds after the application of the conditioning stimulus, the first and second test stimulus (pain pressure thresholds) is measured at the non-affected tibialis anterior muscle. The difference between second and first test stimulus is calculated and used for the analysis.
  Unit of the outcome measure is kilogram per square centimeter (kg/cm2).
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery.
Degree of pain facilitation | Time frame up to 12 months post-surgery
  This measurement is performed using a 26 g monofilament. Repetitive 30 stimuli will be applied at affected lateral trunk. Perceived intensity of stimulus will be assessed between 0 and 10.
  Pain intensity scores are recorded on the Numerical Rating Scale after the first stimuli and after 30 consecutive stimuli (65). Difference between Numerical Rating Scale after 30 stimuli and the first stimulus is calculated and used for the analysis.
  Score is between 0 - 10. Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of altered body perception | Time frame up to 12 months post-surgery
  Body perception is evaluated by the Fremantle Upper Limb Awareness Questionnaire.
  This questionnaire evaluates neglect-like symptoms, reduced sensory acuity, and perceived size at arm and trunk/breast and consists of 9 items. Each item is scored on a 5-point Likert scale from 0 (never) to 4 (always). Higher scores indicate a greater sense of bodily unawareness in the affected arm or trunk/breast.
  Total score ranges between 0 - 63.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery.
Severity of subjective arm lymphedema | Time frame up to 12 months post-surgery
  Severity of subjective arm lymphedema is determined based on the severity of the difference in the size of 3 sites (hand, lower arm, and upper arm) by two items: 1) frequency with "0: not applicable to 4: almost always" and 2) severity with "0: not applicable to 3: very noticeable".
  Total score ranges between 0 and 21.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery
Severity of subjective trunk lymphedema | Time frame up to 12 months post-surgery
  The severity of subjective trunk BCRL will be determined by the severity of the difference in the size of trunk and breast/ breast region by two items: 1) frequency with "0: not applicable to 4: almost always" and 2) severity with "0: not applicable to 3: very noticeable".
  Total score is between 0 and 14.
  Assessment at pre-surgery (baseline) and 1 month, 6 months, and 12 months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- University Hospitals of Leuven, center for lymphedema, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gursen C, Dylke ES, Moloney N, Meeus M, De Vrieze T, Devoogdt N, De Groef A. Self-reported signs and symptoms of secondary upper limb lymphoedema related to breast cancer treatment: Systematic review. Eur J Cancer Care (Engl). 2021 Sep;30(5):e13440. doi: 10.1111/ecc.13440. Epub 2021 Mar 18. PMID 33733550
- [Background] Svensson BJ, Dylke ES, Ward LC, Black DA, Kilbreath SL. Screening for breast cancer-related lymphoedema: self-assessment of symptoms and signs. Support Care Cancer. 2020 Jul;28(7):3073-3080. doi: 10.1007/s00520-019-05083-7. Epub 2019 Oct 22. PMID 31641870
- [Background] De Groef A, Devoogdt N, Gursen C, Moloney N, Warpy V, Daelemans J, Dams L, Haenen V, Van der Gucht E, Heroes AK, De Vrieze T, Dylke E. Correction to: Sensory signs and symptoms in women with self-reported breast cancer-related lymphedema: a case-control study. J Cancer Surviv. 2022 Dec;16(6):1508-1509. doi: 10.1007/s11764-021-01125-4. No abstract available. PMID 34716888
- [Background] Fu MR, Axelrod D, Cleland CM, Qiu Z, Guth AA, Kleinman R, Scagliola J, Haber J. Symptom report in detecting breast cancer-related lymphedema. Breast Cancer (Dove Med Press). 2015 Oct 15;7:345-52. doi: 10.2147/BCTT.S87854. eCollection 2015. PMID 26527899
- [Background] Sackey H, Johansson H, Sandelin K, Liljegren G, MacLean G, Frisell J, Brandberg Y. Self-perceived, but not objective lymphoedema is associated with decreased long-term health-related quality of life after breast cancer surgery. Eur J Surg Oncol. 2015 Apr;41(4):577-84. doi: 10.1016/j.ejso.2014.12.006. Epub 2015 Jan 13. PMID 25659877
- [Background] Terada M, Yoshimura A, Sawaki M, Hattori M, Naomi G, Kotani H, Adachi Y, Iwase M, Kataoka A, Sugino K, Mori M, Horisawa N, Ozaki Y, Iwata H. Patient-reported outcomes and objective assessments with arm measurement and bioimpedance analysis for lymphedema among breast cancer survivors. Breast Cancer Res Treat. 2020 Jan;179(1):91-100. doi: 10.1007/s10549-019-05443-1. Epub 2019 Sep 18. PMID 31535321
- [Background] Sayko O, Pezzin LE, Yen TW, Nattinger AB. Diagnosis and treatment of lymphedema after breast cancer: a population-based study. PM R. 2013 Nov;5(11):915-23. doi: 10.1016/j.pmrj.2013.05.005. Epub 2013 May 17. PMID 23684778
- [Background] McLaughlin SA, Wright MJ, Morris KT, Sampson MR, Brockway JP, Hurley KE, Riedel ER, Van Zee KJ. Prevalence of lymphedema in women with breast cancer 5 years after sentinel lymph node biopsy or axillary dissection: patient perceptions and precautionary behaviors. J Clin Oncol. 2008 Nov 10;26(32):5220-6. doi: 10.1200/JCO.2008.16.3766. Epub 2008 Oct 6. PMID 18838708
- [Derived] Gursen C, Meeus M, Verbeelen K, Vets N, Spincemaille L, Smeets A, Thomis S, Fieuws S, Vanderheyden H, Gebruers N, Tjalma W, Johansson K, Keeley V, De Groef A, Devoogdt N. LymphSens study: the enigma of subjective lymphoedema - how often and why do patients report lymphoedema after breast cancer treatment without an objective measurable swelling? The role of lymphatic and sensory processing problems: a protocol for a multicentre prospective longitudinal study. BMJ Open. 2025 Jun 8;15(6):e099990. doi: 10.1136/bmjopen-2025-099990. PMID 40484423